CLINICAL TRIAL: NCT06494605
Title: Early Neurodivergent Developmental Trajectories in Toddlers and Young Children on the Autism Spectrum and Effectiveness of the Early Start Denver Model in Community Settings
Brief Title: Early Neurodivergent Developmental Trajectories in Autism and in Response to the ESDM Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Istituto Superiore di Sanità (Other); Messina, Italy (Other); Società Cooperativa Sociale AUDACIA (Unknown); Associazione Ulisse (Unknown); La Linea Curva (Unknown)
Responsible Party: Principal Investigator, Liliana Ruta, MD, PhD, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-010
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; early support; children; ESDM; individual trajectories
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental study (Experimental): The experimental group consists of 33 children diagnosed with early signs of neurodivergence or diagnosis of autism. The sample is aged between 18 and 48 months
  Interventions: Behavioral: Early Start Denver Model (ESDM)

INTERVENTIONS:
Behavioral: Early Start Denver Model (ESDM) — The Early Start Denver Model (ESDM) is an early naturalistic and behavioural intervention for children with initial signs of neurodivergence or on the autism spectrum between the ages of 12-48 months. This early intervention aims to increase the rates of development in several domains and to decrease the characteristics of autism conditions that hinder children's ability to learn from everyday experiences and interactions.

SUMMARY:
Early support is thought to be key to ensure a better quality of life for young children on the autism spectrum. Among early support, different evidence-based approaches have combined the principles of developmental and behavioral science within a naturalistic and interactive frame and grouped under the umbrella of Naturalistic Developmental Behavioral Interventions (NDBI). In the context of NDBIs, the Early Start Denver Model is a manualized support that has reported evidence of efficacy for therapist-, group- and caregiver-implemented support, in multiple research as well as community based settings, different countries and languages (Rogers & Dawson, 2010). Understanding the effects of support characteristics and intensity on individual learning has a major impact on the delivery systems organization and policies, sustainability in low resources community settings and to provide the necessary support to the family. However, a direct comparison among different types and intensity of early support in community setting and relatively low access to standardized and intensive programs, have not been adequately explored. For this reason, the aim of this study is to investigate, in a community setting in the Italian context, the impact of ESDM and support intensity on individual developmental trajectories.

ELIGIBILITY:
Inclusion Criteria:

* unimpaired hand use
* parent agreement to have a caregiver present during all home sessions
* attendance at all intake sessions
* permission to videotape evaluations and ESDM treatment
* Italian as one primary language of the parent
* unimpaired hearing and vision
* developmental quotient of 35 or higher on the Griffith Scale
* meets all of these autism spectrum disorder diagnostic criteria through the Autism Diagnostic Observation Schedule (ADOS; cutoff score of 12 if child produces no words or 10 if child produces some words)

Exclusion Criteria:

* serious parental substance abuse
* parental self-report of bipolar disorder or psychosis
* known genetic syndromes
* serious medical conditions (e.g., encephalitis, concussion, seizure disorder)
* significant sensory impairment
* birth weight <1600 grams and/or gestational age < 34 weeks
* history of intraventricular hemorrhage
* known exposure to neurotoxins (including alcohol, drugs)
* non-Italian-speaking parents

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) | The test will be scheduled pre intervention (T0) after six months (T2) and at the study conclusion, 1 year (T4). The complete test takes 90 minutes.
  The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) is the "gold standard" for the assessment of autism spectrum disorder. It is an activity-based assessment evaluating communication skills, social interaction and imaginative use of materials through five modules:
  * Toddler Module: for children from 12 to 30 months who have not yet developed fluent language. It provides a risk indicator.
  * Module 1: for children from 31 months without fluent language. Autism Spectrum: total score ≥ 12 Autism: total score ≥ 16
  * Module 2: for children who produce complete sentences even if not fully fluent, even under 30 months.
  Autism Spectrum: total score ≥ 8 Autism: total score ≥ 12
  * Module 3: for children and young adolescents with fluent verbal language. Autism Spectrum: total score ≥ 7 Autism: total score ≥ 10
  * Module 4: for late adolescents and adults with fluent verbal language. Autism Spectrum: total score ≥ 7 Autism: total score ≥ 10
Griffith Scale Development Scales (GMDS) | The test will be scheduled pre intervention (T0), after three months (T1), after six months (T2), after nine months (T3) and at the study conclusion, 1 year (T4). The complete test takes 90 minutes.
  The Griffith Mental Development Scales (GMDS-ER) assess the developmental quotient of infants and young children from birth to eight years in five developmental areas (Griffith, 2006):
  * Locomotor (gross motor skills including balance, coordination and control movements);
  * Personal Social (personal independence and social development);
  * Hearing and Language (receptive and expressive languages);
  * Eye and Hand Coordination (fine motor skills, manual dexterity and visual monitoring skills);
  * Performance (visuospatial skills, speed of working and precision). Subscale quotients are calculated by dividing the developmental age corresponding to each subscale by the actual chronological age and multiplying by 100.The General Quotient (GQ) and each subscale quotient have a mean of 100 points (Standard Deviation (SD) = 15 points).The GQ raw score is the sum of the subscales raw scores. A GQ or a subscale quotient <70 points (>2SD below the mean) indicates developmental delay.
Vineland Adaptive Behavior Scales (VABS) | The test will be scheduled pre intervention (T0), after three months (T1), after six months (T2), after nine months (T3) and at the study conclusion, 1 year (T4). The complete test takes 60 minutes.
  The Vineland Adaptive Behavior Scales (VABS) is a standardized assessment tool and measure adaptive behavior (Sparrow et al., 2005). It uses standard scores, percentile ranks and v-scale scores to evaluate an individual's performance across different domains: Communication, Daily Living Skills, Socialization, Motor Skills (optional), and Maladaptive Behavior (optional).
  The key metrics include:
  1. Adaptive Behavior Composite (ABC): It is a composite of the domain scores linked to general adaptive functioning.
  2. Domain Scores: The domains are: Communication, Daily Living Skills, Socialization, and optionally, Motor Skills and Maladaptive Behavior.
  3. Subdomain Scores: These subdomain provide more detailed information within each domain.
  The scores are norm-referenced, meaning they compare an individual's performance to a representative sample of the population, with an average (mean) score of 100 and a standard deviation of 15 for the ABC and domain scores.
Early Start Denver Model Curriculum | The test will be scheduled pre intervention (T0), after three months (T1), after six months (T2), after nine months (T3) and at the study conclusion, 1 year (T4). The complete curriculum takes 90 minutes.
  The Early Start Denver Model Curriculum Checklist for Young Children with Autism is used to provide a comprehensive assessment of the skills of toddlers and preschoolers with autism spectrum disorder across a range of developmental domains and to set individualized instructional goals. Administered every 12 weeks, it is an essential tool in the intervention program outlined in Early Start Denver Model for Young Children with Autism manual.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Ruta, Principal Investigator — National Research Council of Italy, Institute for Biomedical Research and Innovation (CNR-IRIB)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB)-National Reasearch Council (CNR),, Messina, ME, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruschetta, R., Campisi, S., Mastrogiuseppe, M., Leonardi, E., Aiello, S., Salvatore, C., ... & Tartarisco, G. (2023, July). A deep learning approach for automatic video coding of deictic gestures in children with autism. In 2023 3rd International Conference on Electrical, Computer, Communications and Mechatronics Engineering (ICECCME) (pp. 1-6). IEEE.
- [Background] Campisi, A., Mastrogiuseppe, M., Aiello, S., Leonardi, E. L. I. S. A., Fama, F. I., Carrozza, C., ... & Ruta, L. (2023). Early Language-Specific Developmental Differences in Young Children with and without Autism. INSAR 2023.
- [Background] Mastrogiuseppe, M., Leonardi, E. L. I. S. A., Aiello, S., Fama, F. I., Campisi, A., Carrozza, C., ... & Ruta, L. (2023). Characteristics of Gesture Communication in Young Children with Autism during Naturalistic Play Interactions. INSAR 2023.
- [Background] Fama, F. I., Aiello, S., Carrozza, C., Leonardi, E. L. I. S. A., Campisi, A., Blandino, C., ... & Ruta, L. (2023). Parental Interaction Style during Naturalistic Play Activities in Young Children with and without Autism. INSAR 2023.
- [Background] Ruta, L., Mastrogiuseppe, M., Fama, F. I., Carrozza, C., Leonardi, E. L. I. S. A., Aiello, S., ... & Pioggia, G. (2023). Early Developmental Trajectories in Response to Early Start Denver Model: Effects of Treatment Type and Intensity in Community Settings. INSAR 2023.